CLINICAL TRIAL: NCT05928195
Title: Acute, Dose-Response Effects of Organic Guayusa Extract on Cognitive Performance, Mood, Resting Metabolism, and Blood Pressure, Heart Rate, and Heart Electrical Activity
Brief Title: Acute Effects of Organic Guayusa Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathaniel Jenkins (Other)
Responsible Party: Sponsor-Investigator, Nathaniel Jenkins, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 202202283
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Acute Physiological Effects of Organic Guayusa Extract
Keywords: dietary supplementation; cognitive performance; metabolism; heart rate; blood pressure; electrocardiogram; mood

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-Dose Guayusa Extract (Experimental): Acute, single dose of 600 mg Organic Guayusa Extract
  Interventions: Dietary Supplement: Acute Moderate-Dose Guayusa Extract Supplementation
- High-Dose Guayusa Extract (Experimental): Acute, single dose of 1200 mg Organic Guayusa Extract
  Interventions: Dietary Supplement: Acute High-Dose Guayusa Extract Supplementation
- Placebo (Placebo Comparator): Acute, single dose of Placebo (dextrose)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Acute Moderate-Dose Guayusa Extract Supplementation — Participants will consume two vegan capsules with one capsule containing 600 mg AmaTea® and 1 containing 600 mg dextrose.
  Arms: Moderate-Dose Guayusa Extract
Dietary Supplement: Acute High-Dose Guayusa Extract Supplementation — Participants will consume two vegan capsules with each capsule containing 600 mg AmaTea® (1200 mg total).
  Arms: High-Dose Guayusa Extract
Dietary Supplement: Placebo — Participants will consume two vegan capsules with each capsule containing 600 mg dextrose (1200 mg total).
  Arms: Placebo

SUMMARY:
Guayusa extract is a caffeinated tea leaf unique blend of antioxidants and caffeine. It is marketed as an ingredient that can help support energy and performance with potential health-related benefits. It has also been indicated as being as safe as any other existing teas (i.e., green tea). However, no studies have previous studied the dose-response effects of guayusa extract for supporting cognitive function, mood, metabolism, nor its effects on resting heart rate, blood pressure, and electrocardiogram characteristics.

DETAILED DESCRIPTION:
Guayusa extract is a caffeinated Amazonian 'super-leaf' belonging to the holly species that contains a unique blend of polyphenol antioxidants and caffeine (~20% caffeine, 30% chlorogenic acids, 5% catechins). It is also remarkably low in tannins which are responsible for the bitter taste found in most teas - giving it a sweet flavor profile. As such, it is marketed as an ingredient that can help support energy and performance (e.g., via caffeine content) with potential health-related benefits due to its antioxidant properties. Indeed, ingredients such as these are often consumed by individuals prior to exercise in order to help improve neurocognitive performance, mood, or otherwise to support health-related goals such as metabolism. Whereas several studies have suggested that caffeine and chlorogenic acid consumption may improve performance, mood, and concentration, and some evidence in animals have linked catechin consumption to improved health outcomes, no studies have previous studied whether guayusa extract supplementation helps to support these, nor has the dose-effectiveness been tested, in humans.

In this study, the effects of acute dietary supplementation with two different doses of botanical organic guayusa extract on neurocognitive/motor-cognitive performance, mood, focus, and jitteriness, resting metabolism, and resting heart rate, blood pressure, and electrocardiogram characteristics will be examined.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years, inclusive
* Physically active (>=150 min/wk or >=75 min/wk Moderate or Vigorous PA) for >=3 months
* BMI <= 30 kg/m2
* Otherwise healthy
* Habitual caffeine consumption >=200 mg/day OR 1-week washout of current caffeine usage prior to participation

Exclusion Criteria:

* Current injury or illness that precludes exercise participation
* Current nicotine or cannabis use
* Use of prescription ADD/ADHD, anti-depressant, or other central acting medication, or previously diagnosed ADD/ADHD, clinically depressed, or generalized anxiety disorder
* Current taking prescription stimulants (i.e., Adderall, Ritalin, Vyvanse, etc.)
* Participants with a history of metabolic, hepatorenal, musculoskeletal, autoimmune, or neurologic disease; or currently taking thyroid, hormonal, hyperlipidemic, hypoglycemic, anti-hypertensive, anti-inflammatory, or anti-coagulant medications.
* Treated for Metabolic Syndrome or having been clinically diagnosed with, or taking medication for a cardiometabolic-disorder (e.g., Pre-diabetes, Type II diabetes, high blood pressure, obesity, hypercholesterolemia, etc.)
* Currently pregnant or lactating
* Diagnosed allergy to any ingredient present within the study treatments
* Current competitive NCAA athlete
* Inability or unwillingness to comply with the controls and conditions of the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-07-13 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Mood | 90-minutes Post-supplementation
  Calculated as Total Mood Disturbance (arbitrary units) using the Profile of Mood States Short Form Questionnaire.
Psychomotor Speed | 60-minutes Post-supplementation
  How well participant perceived, attends, responds to visual-perceptive information, and performs motor speed and fine motor coordination. Calculated as the sum of finger taps in finger tapping test and correct responses in the symbol digit coding test.
Executive Function | 60-minutes Post-supplementation
  How well participant recognized rules, categories, and manages or navigates rapid decisions making. Calculated as the differences between Shifting Attention Test Correct Responses and Errors.

SECONDARY OUTCOMES:
Jitteriness | 90-minutes Post-supplementation
  Participants will describe how jittery they feel after supplemention using a 0-100 mm visual analog scale.
Focus | 90-minutes Post-supplementation
  Participants will describe how focused they feel after supplemention using a 0-100 mm visual analog scale.
Energy | 90-minutes Post-supplementation
  Participants will describe how energetic they feel after supplemention using a 0-100 mm visual analog scale.
Resting Metabolic Rate | 50 minutes post-supplementation
  Resting metabolic rate (kcal/min) will be quantified from resting, fasted analyses of pulmonary gas exchange.
Resting Fat Oxidation | 50 minutes post-supplementation
  Resting fat oxidation (g/min) will be quantified from resting, fasted analyses of pulmonary gas exchange.
Resting Heart Rate | -10 minutes before supplementation, 40 minutes post-supplementation
  Heart rate (bpm) will be quantified from a standard 12-lead ECG
Resting Blood Pressure | -10 minutes before supplementation, 40 minutes post-supplementation
  Systolic, diastolic, and pulse pressures (mmHg) will be quantified from brachial artery via automated sphygmomanometer.
QTc Interval | -10 minutes before supplementation, 40 minutes post-supplementation
  QTc Interval (ms) will be quantified from a standard 12-lead ECG
Motor-Cognitive Reaction Time | 100-minutes Post-supplementation
  Motor-cognitive reaction times (ms) will be quantified from motor cognitive (reactionary hop) tests
Sustained Attention | 60-minutes Post-supplementation
  How well a subject can direct and focus cognitive activity on specific stimuli. Derived from performance on the 4-part continuous performance task test.
Working Memory | 60-minutes Post-supplementation
  How well a subject can perceive and attend to symbols using short-term memory processes.
Cognitive Flexibility | 60-minutes Post-supplementation
  How well subject is able to adapt to rapidly changing and increasingly complex set of directions and/or to manipulate the information. Assessed from the Shifting Attention Task and Stoop Test as the Shifting Attention Task Correct Responses - Shifting Attention Task Incorrect Responses and Stroop Commission Errors.

OTHER OUTCOMES:
Vigor | 90-minutes Post-supplementation
  Vigor will be quantified using the Profile of Mood State Short Form Questionnaire.
Tension | 90-minutes Post-supplementation
  Tension will be quantified using the Profile of Mood State Short Form Questionnaire.
Fatigue | 90-minutes Post-supplementation
  Fatigue will be quantified using the Profile of Mood State Short Form Questionnaire.
Anger | 90-minutes Post-supplementation
  Anger will be quantified using the Profile of Mood State Short Form Questionnaire.
Confusion | 90-minutes Post-supplementation
  Confusion will be quantified using the Profile of Mood State Short Form Questionnaire.
Stress | 90-minutes Post-supplementation
  Stress will be quantified using the Profile of Mood State Short Form Questionnaire.
Composite Memory | 60-minutes Post-supplementation
  How well subject can recognize, remember, and retrieve words and geometric figures. Assessed as a composite performance indicator during the Verbal Memory and Visual Memory Tests.
Reaction Time | 60-minutes Post-supplementation
  How quickly the subject can react, in milliseconds, to a simple and increasingly complex direction set.
Complex Attention | 60-minutes Post-supplementation
  Ability to track and respond to a variety of stimuli over lengthy periods of time and/or perform mental tasks requiring vigilance quickly and accurately.
Reasoning | 60-minutes Post-supplementation
  How well is subject able to recognize, reason and respond to non-verbal visual-abstract stimuli. Assessed from the non-verbal reasoning test as the difference between the number of correct responses and commission errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Laboratory of Applied Physiology and Lifestyle Medicine, Iowa City, Iowa, United States